CLINICAL TRIAL: NCT00342316
Title: Prospective Controlled Clinical Study of Allogeneic Stem Cell Transplantation With Reduced Conditioning (RICT) Versus Best Standard of Care in Acute Myeloid Leukemia (AML)in First Complete Remission (CR)
Brief Title: Reduced Intensity Conditioning Transplantation Versus Standard of Care in Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: The Canadian Blood and Marrow Transplant Group (Network); Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRALG1/02
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Stem Cell Transplantation; Reduced Intensity Conditioning; Survival; Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: Formally, this is not Phase III study, since there are no new drugs or interventions. Rather - a prospective, controlled study where we include pts aimed for alloSCT before any donor search. Both groups of pts (with or without a matched donor) are followed ≥2yrs. The hypothesis is that pts with a donor do better than those without a donor (sib and/or unrelated).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell transplant (RICT) (Experimental): Receiving intervention consisting of Reduced Intensity Conditioning Stem Cell Transplantation
  Interventions: Procedure: Reduced Intensity Conditioning Stem Cell Transplantation
- Control arm (No Intervention): Treatment according to standard of care, i.e. not undergoing RICT

INTERVENTIONS:
Procedure: Reduced Intensity Conditioning Stem Cell Transplantation — One of the following conditioning regimens:
  1. Busulphan (orally or IV), fludarabine
  2. Fludarabine, carmustine, melfalan
  3. Cyclophosphamide, fludarabine
  Arms: Stem cell transplant (RICT)

SUMMARY:
This study compares overall survival between patients with acute myeloid leukemia, who are in complete remission following initial treatment with chemotherapy and whose remission is maintained either with a transplantation of stem cells obtained from a sibling or unrelated donor or with standard treatment, which is additional chemotherapy.

The study hypothesis is that the group transplanted with stem cells from a donor will have a superior survival compared with patients treated with standard of care.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to determine whether RICT leads to an improved overall survival compared to conventional treatment for AML.

The secondary objectives of this study are to determine if:

* RICT leads to a superior long-term overall survival compared to conventional therapy.
* RICT leads to a superior disease-free survival compared to conventional therapy.
* Time to relapse is different between RICT and control groups.
* Quality of life is different between the two treatment groups.
* in RICT patients only:

  * Safety and feasibility of the procedure
  * Incidence and severity of acute and chronic Graft versus Host Disease (GvHD)
  * Rate of complete and partial chimerism

Study Population:

* Newly diagnosed patients with de novo or secondary AML, intermediate or poor risk, in first complete remission aged 51-70 years.
* Not planned for a full-dose allogeneic transplant.
* According to the investigator, fit for a RICT if a suitable donor (sibling or unrelated) is found, and also fit for further consolidation chemotherapy in case no suitable donor is found.

Procedures:

Patients will receive induction therapy according to institutional practice and can be included after achieving complete remission. Patients for whom a full-dose conditioned allogeneic transplantation is planned will not be approached, neither will patients who are for other reasons judged to be ineligible for a RICT. Eligible patients will be informed about the study. After the patient's consent has been obtained, potential sibling donor(s) will be briefly informed about the study and asked if they are willing to undergo HLA-typing. Siblings with evident contraindications to granulocyte colony stimulating factor (G-CSF) or collection of peripheral blood stem cells should not proceed to HLA-typing. A search for an unrelated matched donor (MUD) will be initiated if there is no potential sibling donor, or if sibs are not HLA-identical or otherwise not fit for the donation procedure. A patient's inclusion in the study is when blood sampling for tissue typing (HLA-typing) of the first potential sibling donor is made, or when a search warrant for a MUD is dispatched.

* Note: To enable an early donor search, patients may be registered, but not included, for the study prior to CR. These patients will be included at date of achieved CR. Registered patients not achieving CR will not be included.

Included patients with a HLA-identical sibling or with an identified MUD will be assigned to the RICT group, and included patients without such a donor will automatically be in the control group. This is a HLA-based assignment, and the final intent-to-treat analysis will be based on the treatment assignment.

After treatment assignment, patients on the control arm should receive consolidation therapy as per institutional practice, whereas patients on the RICT arm may proceed directly to RICT or receive one or maximum two consolidation courses. Patients should be in complete remission at the time of transplant. All patients will be followed for relapse and survival for a period of at least three years.

The inclusion of 352 patients in complete remission provides a statistical power of 90 % to detect a difference in overall survival at three years of 20 percentage points, ie from 30 % of control patients to 50 % in RICT patients.

Inclusion was terminated 2016-07-19 after 360 registered patients. However, some pts were excluded due to grave protocol deviations or withdrawn consent. The data base was locked in June 2018 for analysis with 309 pts (after exclusions). Follow-up was >2 yrs fo all pts.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with de novo or secondary AML
* Intermediate or poor risk
* In first complete remission
* Age 51-70 years
* Fit for the procedure
* Fit for further consolidation chemotherapy

Exclusion Criteria:

* Planned for a full-dose allogeneic transplant

Ages: 51 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2003-12-18; Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From Inclusion until one of the above events (≥2yrs in all surviving pts).
  OS is the time from Inclusion to death, lost to follow-up, refusal, or study termination.

SECONDARY OUTCOMES:
Disease-free survival | From Inclusion to relapse, death or study termination. Follow-up ≥24 mo in all surviving pts.
  DFS is the time from Inclusion until date of first documented relapse, death from any cause whichever came first, assessed until study termination.
Quality of Life for pts in the RICT and Control Groups. | All pts were asked to fill out the instrument at 12 and 24 months after inclusion
  European Organization for Research and Treatment of Cancer (EORTC). Quality of Life Questionnaire (QLQ), Cancer C) #30. An instrument commonly used for the evaluation of QoL after under and after cancer treatment
Non-relapse mortality (NRM). Numbers and causes of death in non-relapsed pts | From Inclusion to relapse or death until study termination.
  NRM is death without preceding relapse, from Inclusion to study termination.
Acute and Chronic Graft-versus-Host Disease (GvHD) | Acute GvHD: From transplant to 3 months. Chronic From transplantation to relapse, death or study termination
  In transplanted pts only. Acute GvHD appears from transplant to 100 days. Chronic GvHD occurs later, and often remains for years. Both are clinical diagnoses and cGvHD grading were performed annually until death or study termination.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Brune, MD, PhD, Principal Investigator — Göteborg University
Locations (25):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austalasian Leukaemia &Lymphoma Group Limited, East Melbourne, Victoria
- Canada (8):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - McMaster Site Ward 3Z, Hamilton Health Sciences, Hamilton, Ontario
  - Hematology, Ottawa Hospital, Ottawa, Ontario
  - Hématologie, Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hematology, Royal Victoria Hospital, Montreal, Quebec
  - Hématologie, Hospital CHA Enfant-Jésus, Québec, Quebec
  - L'Hôtel Dieu de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Tartu University Hospital, Tartu, Estonia
- Turku University Hospital, Turku, Finland
- Dept of Hematology, University Hospital, Freiburg im Breisgau, Germany
- University Hospital of Patras, Pátrai, Greece
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington
- Section of Hematology, National Hospital, Oslo, Norway
- Sweden (7):
  - Department of Hematology, Sahlgrenska University Hospital, Gothenburg
  - Sunderby Hospital, Luleå
  - Skåne University Hospital Lund, Lund
  - University Hospital Örebro, Örebro
  - Karolinska University Hospital Huddinge, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Uppsala Akademiska Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No